CLINICAL TRIAL: NCT01690286
Title: An Open-Label Study to Assess the Effects of Repeated Twice-Daily Doses of Ketoconazole on the Steady-State Pharmacokinetics of JNJ-38518168 in Healthy Subjects
Brief Title: Effect of Ketoconazole on the Pharmacokinetics of JNJ-38518168 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100915; 38518168ARA1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2012-09-19; First posted 2012-09-21 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Healthy
Keywords: Healthy; Ketoconazole; JNJ-38518168; Pharmacokinetics
MeSH Terms: interventions — Ketoconazole

ARMS (3):
- Group 1: JNJ-38518168 3 mg/ ketoconazole (Experimental)
  Interventions: Drug: JNJ-38518168 3 mg; Drug: Ketoconazole 200 mg
- Group 2: JNJ-38518168 30 mg/ ketoconazole (Experimental)
  Interventions: Drug: JNJ-38518168 30 mg; Drug: Ketoconazole 200 mg
- Group 3: JNJ-38518168 10 mg/ ketoconazole (optional) (Experimental)
  Interventions: Drug: JNJ-38518168 10 mg; Drug: Ketoconazole 200 mg

INTERVENTIONS:
Drug: JNJ-38518168 3 mg — One oral daily dose of JNJ-38518168 3 mg for 25 days.
  Arms: Group 1: JNJ-38518168 3 mg/ ketoconazole
Drug: JNJ-38518168 30 mg — One oral daily dose of JNJ-38518168 30 mg for 25 days.
  Arms: Group 2: JNJ-38518168 30 mg/ ketoconazole
Drug: JNJ-38518168 10 mg — One oral daily dose of JNJ-38518168 10 mg for 25 days.
  Arms: Group 3: JNJ-38518168 10 mg/ ketoconazole (optional)
Drug: Ketoconazole 200 mg — Oral doses of ketoconazole 200 mg every 12 hours, from Day 22 through Day 25.

SUMMARY:
The purpose of this study is to evaluate the effects of repeated twice-daily administration of 200 mg ketoconazole on the steady-state pharmacokinetics of JNJ-38518168.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-sequence, randomized (dose of JNJ-38518168 (3 mg or 30 mg) is assigned by chance), single-center, multiple-dose study designed to assess the potential effects of multiple oral administration of ketoconazole (KTZ) on the steady-state (a situation where the overall intake of a drug is in equilibrium with its elimination) pharmacokinetics of JNJ-38518168. Pharmacokinetics (PK) explores how the drug is absorbed in the body, distributed within the body, and how it is removed from the body over time. The study consists of 3 phases: a Screening Phase of approximately 3 weeks (Days -22 to -2); an Open-Label Phase (Days -1 to 26); and a Follow-up Phase occurring from 7 to 10 days after the last dose of study drug. Participants will be randomly assigned to receive either a daily dose of 3 mg JNJ-38518168 (Group 1) or a daily dose of 30 mg JNJ-38518168 (Group 2) orally administered for 25 days. All participants will receive multiple oral doses of KTZ (200 mg every 12 hours for both Groups 1 and 2) from Day 22 through Day 25. An optional group of participants receiving 10 mg once daily of JNJ-38518168 (Group 3) may be evaluated if the data from Groups 1 and 2 do not allow the sponsor to estimate sufficiently the interaction between KTZ and daily dose of 10 mg JNJ-38518168. The participants will receive an oral dose of the study drugs in the morning of specified days, after an overnight fast for at least 10 hours. Blood samples will be collected at various times throughout the study for evaluation of drug concentrations in plasma. Safety will be assessed by reporting of adverse events, vital signs, physical examination results, weight, and electrocardiogram (ECG) evaluations. Participants will leave the study center on Day 26 after the collection of the last scheduled PK blood sample. For each participant, a follow-up visit will occur 7 to 10 days after the last dose of study drug. For each participant, the total duration of the study is approximately 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent document indicating that the participant understands the purpose of and procedures required for the study and is willing to participate in the study
* If a woman, must be postmenopausal, surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control before, throughout, and for 3 months after the study
* If a man, must agree to use an adequate contraception method, or partner using effective contraception, and to not donate sperm during the study and for 3 months after the study
* Body mass index (BMI; weight [kg]/height2 [m]2) between 18 and 30 kg/m2 (inclusive), and body weight not less than 50 kg
* Blood pressure between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic
* Non-smoker

Exclusion Criteria:

* History of or current clinically significant medical illness, condition or disease that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal lab results at screening or at admission to the study center
* Clinically significant abnormal physical examination or electrocardiogram (ECG) at screening or at admission to the study center
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen and oral contraceptives and hormonal replacement therapy within 14 days before the first dose of study drug is scheduled
* Has a history of malignancy (the tendency of a medical condition, especially tumors, to become progressively worse) within the previous 5 years before screening (certain less serious malignancies during the previous 5 years, such as basal cell carcinoma of the skin which has been adequately treated, may be allowed by the study doctor)
* Donated blood or had a substantial loss of blood within 3 months before first administration of study drug
* Pregnant or currently breast-feeding
* Smoking or using nicotine-containing products within 3 months of screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The plasma concentrations of JNJ-38518168 | From Day 13 up to Day 26
The plasma concentrations of ketoconazole | Day 25

SECONDARY OUTCOMES:
The time to attain steady-state pharmacokinetics following JNJ-38518168 once daily doses for 21 consecutive days | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Neptune City, New Jersey, United States